CLINICAL TRIAL: NCT02322216
Title: A Comparative Study of Olopatadine Hydrochloride Ophthalmic Solution 0.2% QD vs Olopatadine Hydrochloride Ophthalmic Solution 0.1% BID in the Treatment of Allergic Conjunctivitis in Chinese Subjects
Brief Title: Olopatadine Hydrochloride Ophthalmic Solution Study in Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-12-010 (EXC458-C001); 2016-004317-27 (EudraCT Number)
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergies; Ocular
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PATADAY (Experimental): Olopatadine hydrochloride ophthalmic solution 0.2% in the morning and olopatadine 0.2% vehicle in the evening, 1 drop in each eye for 14 days
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution 0.2%; Drug: Olopatadine 0.2% Vehicle
- PATANOL (Active Comparator): Olopatadine hydrochloride ophthalmic solution 0.1%, 1 drop in each eye in the morning and evening, for 14 days
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution 0.1%

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Ophthalmic Solution 0.2%
  Other Names: PATADAY®
  Arms: PATADAY
Drug: Olopatadine Hydrochloride Ophthalmic Solution 0.1%
  Other Names: PATANOL®
  Arms: PATANOL
Drug: Olopatadine 0.2% Vehicle — Inactive ingredients used as placebo comparator
  Arms: PATADAY

SUMMARY:
The purpose of this study is to evaluate olopatadine 0.2% QD (once per day) compared to olopatadine 0.1% BID (twice per day) in the treatment of ocular itching associated with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity;
* History of allergic conjunctivitis within the last 2 years;
* Positive skin prick test or skin intradermal test documented by a lab report within 24 months of, or at the baseline visit;
* Clinical diagnosis of allergic conjunctivitis with specific signs and symptoms;
* Understand and sign an informed consent form;
* Willing and able to make required study visits and follow study instructions, and comply with dosing study medication as instructed;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Contraindications or hypersensitivity to study medications or their components;
* Best-corrected visual acuity (BCVA) score worse than 55 ETDRS letters (equivalent to approximately 0.60 logMAR, 20/80 Snellen, or 0.25 decimal) in either eye;
* Any ocular condition that could affect the study outcomes;
* Presumed or actual ocular infection or history of ocular herpes in either eye;
* Known history of retinal detachment, diabetic retinopathy, or any progressive retinal disease;
* Willing and able to avoid the use of any other topical ocular medication(s) (including artificial tear products);
* Any significant illness that could be expected to interfere with the study, particularly any autoimmune disease;
* Intraocular surgery in either eye within 6 months, or ocular laser surgery in either eye within 3 months, or anticipation of ocular surgery during the study; ocular trauma in either eye within 3 months of baseline visit;
* Clinically relevant recent (within 6 months of baseline visit) history of or current severe, unstable, or uncontrolled cardiovascular, pulmonary, hepatic, renal, autoimmune disease and other relevant systemic diseases that would preclude the safe administration of a topical antihistamine/mast cell stabilizer in the opinion of the Investigator;
* Use of systemic medication(s) on a chronic dosing regimen for less than 1 month or have changed dosage within the month prior to baseline visit;
* Use of any disallowed medication (topical, topical ophthalmic, systemic and/or injectable) during the period indicated prior to baseline visit. These medications are also not allowed during the study. Disallowed medications include all anti-allergy therapies including those contained in prescription or over-the-counter sleeping aids;
* Use of cold compresses on the eyes during the course of the study;
* Cannot be dosed in both eyes;
* Cannot avoid contact lens wear during the course of the study;
* Therapy with another investigational agent within 30 days of baseline visit, or during the study;
* Women of childbearing potential who are pregnant, intend to become pregnant during the study period, breast-feeding, or not using adequate birth control methods;
* Other protocol-specified exclusion criteria may apply.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Master, Clinical Medicine, Study Director — Alcon (China) Ophthalmic Product Co., Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 study centers located in China.
Pre-assignment Details: Of the 383 enrolled, 130 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (253).
Period: Overall Study
Arm/Group | PATADAY | PATANOL
Started | 126 | 127
Treated (Safety Set) | 126 | 126
Per Protocol Set (PPS) | 123 | 122
Completed | 124 | 123
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who were randomized, received drug, had at least one on-therapy visit, satisfied inclusion/exclusion criteria, and had no major protocol deviations (Per Protocol Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | PATADAY | PATANOL | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (13.72) | 31.9 (12.79) | 32.2 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 86 | 167
  Male | 42 | 36 | 78
Itching Score [Mean (Standard Deviation); unit: units on a scale] — Ocular itching was assessed by the participant on a scale from 0-4, where 0=None and 4=Incapacitating itch.
  units on a scale | 3.35 (0.377) | 3.43 (0.373) | 3.39 (0.376)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worst Ocular Itching Score During the 24 Hours Prior at Day 14
Description: Severity of ocular itching was evaluated as the worst score observed in the past 24 hours prior to each study visit. Ocular itching was assessed by the participant on a scale from 0-4, where 0=None and 4=Incapacitating itch. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 14
Population: Per Protocol Set with non-missing data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | PATADAY | PATANOL
Number analyzed (Participants) | 118 | 112
units on a scale | -2.57 (0.090) | -2.62 (0.092)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of informed consent and for the duration of participation in the study (2 weeks). This analysis group includes all participants who received study treatment. Ocular adverse events are presented for both study eye and non-study eye combined. AEs are reported as pre-treatment and treatment-emergent.
Description: An AE is defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Reports of AEs were obtained through solicited and spontaneous comments from the participants.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- PATADAY: All subjects treated with olopatadine hydrochloride ophthalmic solution 0.2%
- PATANOL: All subjects treated with olopatadine hydrochloride ophthalmic solution 0.1%
Arm/Group | Pre-treatment | PATADAY | PATANOL
Serious Adverse Events (participants affected / at risk) | 0/383 | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 0/383 | 0/126 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.